CLINICAL TRIAL: NCT06876753
Title: Regional Lymph Node Metastasis and Survival Outcomes in Advanced Hepatocellular Carcinoma Receiving Transarterial Chemoembolization and PD-(L)1 Inhibitors-based Immunotherapy
Brief Title: Regional Lymph Node Metastasis and Survival Outcomes in Advanced HCC
Acronym: CHANCE2421
Status: Recruiting | Type: Observational
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, President, Zhongda Hospital
Other Study IDs: CHANCE2421
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: hepatocellular carcinoma; lymph node metastasis; transarterial chemoembolization; immune checkpoint inhibitors; molecular target therapies
MeSH Terms: conditions — Carcinoma, Hepatocellular; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Tumor-draining lymph nodes play an important role in anti-tumor immune responses. In patients with hepatocellular carcinoma (HCC), however, the relationship between regional lymph node metastasis (LNM) and immunotherapy-based efficacy is unclear. This study aimed to evaluate whether extrahepatic LNM is associated with worse survival outcomes as compared to other metastatic sites in patients with advanced HCC.

DETAILED DESCRIPTION:
In patients with advanced-stage hepatocellular carcinoma (HCC), previous studies showed that transarterial chemoembolization (TACE) in combination with immune checkpoint inhibitors (ICIs) and molecular target therapies exhibited better efficacy (PFS and OS) as compared to the ICIs and molecular target therapies. Besides, previous studies showed that tumor-draining lymph nodes play an important role in anti-tumor immune responses in vivo and in vitro studies. However, the relationship between regional lymph node metastasis (LNM) and immunotherapy-based efficacy is unclear. Therefore, this study aimed to evaluate whether extrahepatic LNM is associated with worse survival outcomes as compared to other metastatic sites in patients with advanced HCC who received transarterial chemoembolization (TACE) in combination with ICIs and molecular target therapies. This real-world study may provide further information on treatment selection for clinical practice and trials.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of HCC confirmed by radiology, histology, or cytology;
2. Barcelona Clinic Liver Cancer (BCLC) stage C with the presence of extrahepatic spread;
3. Has not received any previous systemic therapy for HCC (including chemotherapy, molecularly targeted therapy, immunotherapy);
4. Both PD-1/PD-L1 inhibitors and anti-angiogenesis drugs patients received only include marketed drugs but are not limited to HCC approval;
5. TACE was performed after the first PD-1/PD-L1 inhibitor/anti-angiogenic drug treatment or before treatment (within 3 months);
6. Received at least 1 cycle of PD-1/PD-L1 inhibitor/anti-angiogenic drug combination therapy after TACE treatment;
7. Has repeated measurable intrahepatic lesions;

Exclusion Criteria:

1. Cholangiocarcinoma, fibrolamellar, sarcomatoid hepatocellular carcinoma, and mixed hepatocellular/cholangiocarcinoma subtypes(confirmed by histology, or pathology) are not eligible;
2. Unable to meet criteria of combination timeframe described above;
3. Child-Pugh C or PS > 2 or Severe hepatic encephalopathy

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic HCC who received TACE in combination with PD-1/PD-L1 inhibitors and molecular target therapies under real-world practice conditions
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival(OS) | up to approximately 2 years
  OS is defined as the time from the initiation of any combination treatment to death due to any cause.

SECONDARY OUTCOMES:
Progression free survival(PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | up to approximately 2 years
  The PFS is defined as the time from the initiation of any combination treatment to the first documented progressive disease (according to RECIST 1.1) or death due to any cause, whichever occurs first.
PFS per Modified Response Evaluation Criteria in Solid Tumors (mRECIST) | up to approximately 2 years
  PFS is defined as the time from the initiation of any combination treatment to the first documented progressive disease (according to mRECIST) or death due to any cause, whichever occurs first.
Objective response rate(ORR) per RESCIST 1.1 | up to approximately 2 years
  ORR is defined as the proportion of patients with a documented complete response(CR) or partial response(PR) per RECIST 1.1.
ORR per mRECIST | up to approximately 2 years
  ORR is defined as the proportion of patients with a documented CR or PR per mRECIST.
Disease Control Rate (DCR) per RESCIST 1.1 | up to approximately 2 years
  DCR is defined as the percentage of participants who have a best overall response of CR, PR, or stable disease (SD)per RESCIST 1.1.
DCR per mRECIST | up to approximately 2 years
  DCR is defined as the percentage of participants who have a best overall response of CR, PR, or stable disease (SD) per mRECIST.
Duration of Response (DOR) per RESCIST 1.1 | up to approximately 2 years
  DOR is determined by disease assessment and is defined as the time from the first documented evidence of a response of CR or PR until the first documented disease progression (according to RESCIST 1.1) or death due to any cause, whichever occurs first.
DOR per mRECIST | up to approximately 2 years
  DOR is determined by disease assessment and is defined as the time from the first documented evidence of a response of CR or PR until the first documented disease progression (according to mRECIST) or death due to any cause, whichever occurs first.
Adverse event(AE) per Common Terminology Criteria for Adverse Events(CTCAE) 5.0 | up to approximately 2 years
  The percentage and degree of patients who experience at least one AE, whether or not considered related to the treatment, according to CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Gao-jun Teng, M.D, Principal Investigator — Zhongda hospital, Southeast university, Nanjing, China
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China